CLINICAL TRIAL: NCT04564196
Title: Feasibility Study of the Collection of the Breath Metabolome From Healthy Parturients During Labor
Brief Title: Breath Metabolomics in the Laboring Parturient
Status: Terminated | Type: Observational
Why Stopped: Staffing and equipment complications have paused further enrollment until resolved
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cedar J. Fowler, M.D. / Ph.D / MPH, Clinical Assistant Professor, Stanford University
Other Study IDs: 54731
Record Dates: First submitted 2020-09-17; First posted 2020-09-25 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Labor Onset and Length Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Induction of Labor: Samples collected from women who present for induction of labor.
  - The parturient will be asked to breathe 2 tidal volume breaths into a single breath collection bag. The breath collection bag will be closed between each breath. The combined 2 tidal volume breaths will count as a single sample.
  Samples will be collected at the following time points for patients presenting for induction of labor:
  A) Baseline: At presentation to labor and delivery unit and prior to initiation of augmentation of labor. A total of 1 sample.
  B) End of 1st stage of labor: At complete cervix dilatation and prior to starting to push. A total of 1 sample will be taken.
  C) End of 3rd stage of labor: Immediately (within 30 minutes) of delivery of the neonate. A total of 1 sample will be taken.
  Interventions: Procedure: Breath Sample
- Spontaneous Labor: Samples will be collected from women who present in spontaneous labor
  - The parturient will be asked to breathe 2 tidal volume breaths into a single breath collection bag. The breath collection bag will be closed between each breath. The combined 2 tidal volume breaths will count as a single sample.
  Samples will be taken at the following endpoints:
  A) End of 1st stage of labor: At completely cervix dilated and prior starting pushing. A total of 1 sample will be taken.
  B) End of 3rd stage of labor: Immediately (within 30 minutes) of delivery of the neonate. A total of 1 sample will be taken.
  Interventions: Procedure: Breath Sample

INTERVENTIONS:
Procedure: Breath Sample — breathe 2 tidal volume breaths into a single breath collection bag. The breath collection bag will be closed between each breath. The combined 2 tidal volume breaths will count as a single sample.

SUMMARY:
This is primarily a feasibility study to determine whether quantitative measurement of volatile organic compounds (VOCs) in the breath of parturients undergoing labor is possible.

Aim A: To determine baseline values of breath metabolites and volatile organic compounds (VOCs) in the breath for term pregnant women.

Aim B: To gather preliminary data to determine breath metabolite and volatile organic compound (VOCs) signature change during labor and delivery.

Aim C: Compare the breath metabolite and volatile organic compound (VOCs) signature women undergoing induction compared to spontaneous vaginal deliveries.

DETAILED DESCRIPTION:
Breath metabolites, also known as volatile organic compounds (VOC's) are produced during periods of increased stress and as a marker of underlying medical conditions. The goal of this project is to collect VOCs within the breath in the initial stages of delivery in otherwise healthy parturients undergoing induction of labor. In addition to a panel of metabolites, we will obtain information on the 3400 compounds which compose the breath metabolome by gas mass spectrometry technology. This is the first step of a larger planned project to develop specialized panels of breath signatures during labor and delivery in parturients.

We will collect breath samples at bedside and measure metabolites in the laboratory. This is a feasibility study which we will use to determine normal values for a term parturient and changes of VOCs during the course of labor. We will also use this data to construct a power analysis and perform a follow-up study to test whether VOCs are associated with different aspects of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy nulliparous women with singleton term (37-41 weeks) pregnant at least 18 years of age.
* Presenting for labor (induction of labor and spontaneous labor) at LPHC.

Exclusion Criteria:

* Participants unable to or refuse to give informed consent
* Participants that do not understand English or are hearing impaired
* Medical History: Chronic disease (HTN, diabetes, asthma)
* Obstetric History during this pregnancy: gestational diabetes, gestational hypertension, pre-eclampsia, Eclampsia
* Multiple gestation
* Any significant fetal anomalies
* Morbid obesity (BMI>50)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with presenting for labor at Stanford.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Profile of volatile organic compounds of the breath | Up to 24 hours
  Mass spectrometry analysis of volatile organic compounds of the breath

CONTACTS AND LOCATIONS:
Overall Officials: Cedar J Fowler, MD/PhD/MPH, Principal Investigator — Stanford University; Pervez Sultan, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after publication and deidentification (text, tables, figures, and appendices). The data will be available for individual participant data meta-analysis.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 24 months following article publication
Access Criteria: Proposals may be submitted up to 24 months following article publication. These proposals will be only reviewed if those investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. After 24 months, the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link to be provided later, please contact PI if unable to locate link).

REFERENCES:
- [Background] Rattray NJ, Hamrang Z, Trivedi DK, Goodacre R, Fowler SJ. Taking your breath away: metabolomics breathes life in to personalized medicine. Trends Biotechnol. 2014 Oct;32(10):538-48. doi: 10.1016/j.tibtech.2014.08.003. Epub 2014 Aug 29. PMID 25179940
- [Background] Norwitz ER, Bonney EA, Snegovskikh VV, Williams MA, Phillippe M, Park JS, Abrahams VM. Molecular Regulation of Parturition: The Role of the Decidual Clock. Cold Spring Harb Perspect Med. 2015 Apr 27;5(11):a023143. doi: 10.1101/cshperspect.a023143. PMID 25918180
- [Background] McLoughlin G. Interventions during pregnancy to prevent preterm birth: An overview of Cochrane systematic reviews. Res Nurs Health. 2020 Apr;43(2):206-207. doi: 10.1002/nur.22005. Epub 2019 Dec 20. No abstract available. PMID 31859369
- [Background] Wallace MAG, Pleil JD. Evolution of clinical and environmental health applications of exhaled breath research: Review of methods and instrumentation for gas-phase, condensate, and aerosols. Anal Chim Acta. 2018 Sep 18;1024:18-38. doi: 10.1016/j.aca.2018.01.069. Epub 2018 Feb 9. PMID 29776545
- [Background] Sukul P, Schubert JK, Trefz P, Miekisch W. Natural menstrual rhythm and oral contraception diversely affect exhaled breath compositions. Sci Rep. 2018 Jul 18;8(1):10838. doi: 10.1038/s41598-018-29221-z. PMID 30022081
- [Background] Nakhleh MK, Haick H, Humbert M, Cohen-Kaminsky S. Volatolomics of breath as an emerging frontier in pulmonary arterial hypertension. Eur Respir J. 2017 Feb 23;49(2):1601897. doi: 10.1183/13993003.01897-2016. Print 2017 Feb. PMID 28232412
- [Background] Cristescu SM, Kiss R, Hekkert St, Dalby M, Harren FJ, Risby TH, Marczin N; Harefield BIOSTRESS study investigators. Real-time monitoring of endogenous lipid peroxidation by exhaled ethylene in patients undergoing cardiac surgery. Am J Physiol Lung Cell Mol Physiol. 2014 Oct 1;307(7):L509-15. doi: 10.1152/ajplung.00168.2014. Epub 2014 Aug 15. PMID 25128523
- [Derived] Hengelage J, Fowler C, Goldsberry MD, Stockert E, Bekemeyer Z, Lee H, Wagner NM, Sultan P, Carvalho B, Gross ER. Quantification of breath metabolites in labouring versus non-labouring patients: a feasibility study. Br J Anaesth. 2025 Nov;135(5):1373-1375. doi: 10.1016/j.bja.2025.07.081. Epub 2025 Sep 9. PMID 40930875